CLINICAL TRIAL: NCT03083574
Title: A Phase II Study to Assess the Safety and the Efficacy of Extracorporeal Photopheresis Using the Theraflex ECP™ for Patients With Refractory Chronic Graft Versus Host Disease (cGVHD)
Brief Title: Extracorporeal Photopheresis Using Theraflex ECP™ for Patients With Refractory Chronic Graft Versus Host Disease (cGVHD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jules Bordet Institute (Other)
Collaborators: Macopharma (Other); Belgian Hematological Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-TC-11
Record Dates: First submitted 2015-01-14; First posted 2017-03-20 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Refractory Chronic Graft Versus Host Disease (cGVHD)
Keywords: Hematology; Chronic graft versus host disease (cGVHD); Extracorporeal photopheresis; Hematopoietic stem cell transplantation; Donor lymphocyte infusion
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Photopheresis Theraflex ECP™ (Experimental): All patients will initially be treated by 6 cycles of extracorporeal photopheresis (i.e. extracorporeal photopheresis on two consecutive days) administered every 2 weeks. Patients will then be evaluated after 3 months and treatment continuation will be decided based on response.
  Interventions: Device: Photopheresis Theraflex ECP™

INTERVENTIONS:
Device: Photopheresis Theraflex ECP™ — The Macopharma (Theraflex ECP™) approach is based on a multistep procedure involving (1) standard mononuclear cell apheresis, (2) injection of the 8-Mop in the apheresis bag, (3) UVA exposure of the bag in the Macogenic illumination device, and (4) reinfusion of the cells into the patients.

SUMMARY:
The present project is a prospective, multicenter, non-randomized, phase II trial which aims to evaluate the clinical impact and the safety of extracorporeal photopheresis (ECP) using the Theraflex system in patients with refractory chronic graft versus host disease (cGVHD) after any type of hematopoietic stem cell transplantation or after donor lymphocyte infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have chronic GVHD (cGVHD) occurring after any type of HSC transplantation : with any type of donor (HLA-identical siblings or HLA-matched or mismatched family or unrelated donor); with any type of conditioning (full-intensity, reduced-intensity, nonmyeloablative, no conditioning); with any type of HSC (bone marrow, PBSC, cord blood) or after donor lymphocyte infusion.
* Patients must have cGVHD primarily affecting at least one of the following organs: skin; oral mucosal; eye; liver; lung; joints; fascia. Gastro-intetinal (GI) cGVHD alone is not a sufficient inclusion criterion.
* Patients must have cGVHD that has already been treated with first-line systemic therapy for at least 1 month at effective doses. First-line systemic therapy must have included at least prednisolone 1 mg/kg/day or equivalent. In case of formal contraindication to steroid therapy, first-line systemic therapy must have included therapeutic doses of at least one of the following drugs: tacrolimus or ciclosporine (if patient not treated with a calcineurin inhibitor at onset of cGVHD), sirolimus, everolimus, mycophenolate mofetyl.
* Patients must require further salvage therapy for cGVHD because of either refractoriness or contraindication/intolerance to current therapy.

Need for salvage therapy is defined by any of the following criteria :

* the development of 1 or more new sites of disease while being treated for chronic GVHD
* progression of existing sites of disease while receiving treatment for chronic GVHD
* failure to improve despite at least 1 month of standard treatment for chronic GVHD,
* relapse/progression of cGVHD while tapering current treatment for cGVHD.

  * Patients may have received any number of previous lines of treatment for cGVHD.
  * Concomitant treatment with other immunosuppressors is allowed if they were started and maintained at constant dosage for at least one month before the start of ECP. Shorter delay can be accepted for patients with highly progressive GVHD requiring salvage therapy.
  * Signed informed consent.
  * Any age.
  * Weight > 15 Kg (because of leukapheresis). Weight <15 Kg is acceptable if a suitable method of leukapheresis has been developed and approved at site.

Exclusion Criteria:

* Patient has received any investigational agent for chronic GVHD in the past 4 weeks.
* Patient has started a new line of systemic therapy for cGVHD in the past 4 weeks. Shorter delay can be accepted for patients with highly progressive GVHD requiring salvage therapy.
* Known sensitivity to psoralen compounds such as 8-methoxypsoralen
* Comorbidities that may result in photosensitivity (coexisting skin cancer or photosensitive disease (such as porphyria, lupus, albinism…)
* Aphakia. MOP is contraindicated in patients with aphakia, because of the significantly increased risk of retinal damage due to the absence of lenses
* Known allergy to one of the components used in apheresis (e.g., heparin and citrate).
* History of heparin-induced thrombocytopenia or patients with serious coagulation disorders.
* Unable to tolerate the apheresis procedure including extracorporeal volume shifts because of uncompensated congestive heart failure, pulmonary edema, severe lung disease, severe renal failure, hepatic encephalopathy, or any other reason.
* Bilirubin > 25 mg/L.
* Absolute neutrophil count < 1.0 x 109 / L despite use of growth factors
* Platelet count < 20 x 109 / L despite platelet transfusion
* HIV seropositivity.
* Uncontrolled infection
* Relapse or progression of the hematological malignancy.
* Eastern Cooperative Oncology Group (ECOG) score > 2.
* Pregnancy or breastfeeding
* Patient is a fertile man or woman who is unwilling to use contraceptive techniques during and for 12 months following treatment.
* Any serious illness with expected survival less than 6 months.
* Any clinically significant medical or other condition that in the investigator's opinion could interfere with the administration of photopheresis or interpretation of study results, or compromise the safety or wellbeing of the patient.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Response rates of chronic GVHD to the Theraflex ECP treatment. | During the study (8 years and 2months)
  Percentage of patients reaching complete response, percentage of patients reaching partial response.
Duration of response. | During the study (8 years and 2months)
  Time from achieving at least a partial response to the time of progression.
GVHD-partial response survival. | During the study (8 years and 2months)
  Time from partial response to either the first progression of GVHD or the date of death, whichever occurs first.
GVHD-free Interval. | During the study (8 years and 2months)
  Interval from the date of complete response to the date of the first progression of GVHD.
GVHD-free survival. | During the study (8 years and 2months)
  Time fromcomplete response to either the first progression of GVHD or the date of death, whichever occurs first.

SECONDARY OUTCOMES:
Percentage of steroid dose saving. | During the study (8 years and 2months)
  Percentage of dose reduction from the date of first ECP to the lowest dose of steroids taken by the patient during a minimum of 3 months (except in case of dose reduction due to adverse events related to steroids)
Discontinuation of immunosuppressive drugs during the ECP treatment | During the study (8 years and 2months)
Occurrence of adverse events and serious adverse events related to extracorporeal photopheresis. | During the study (1 year of follow up after the last treatment)
Incidence of viral, bacterial, fungal and parasitic infections | During the study (8 years and 2months)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lewalle, MD, PhD, Principal Investigator — Jules Bordet Institute
Locations (8):
- Belgium (8):
  - CHU Liège, Liège, Liège
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis Brussel, Jette
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert